CLINICAL TRIAL: NCT05109286
Title: MedXFit Intervention for Predominantly Seated People
Brief Title: A Controlled Trial to Evaluate the Benefits of CrossFit in People Who Work Predominantly in a Sedentary Manner.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Bundeswehr University Munich (Other)
Collaborators: CrossFit Kokoro (Unknown)
Responsible Party: Principal Investigator, Dr. Annette Schmidt, Professor for Sports Biology, Bundeswehr University Munich
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MedXFit
Record Dates: First submitted 2021-10-14; First posted 2021-11-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: People With Predominantly Sedentary Work

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CrossFit training (Experimental): CrossFit training twice a week.
  Interventions: Behavioral: CrossFit
- Control arm (No Intervention): Exercise according to their ideas.

INTERVENTIONS:
Behavioral: CrossFit — CrossFit training
  Arms: CrossFit training

SUMMARY:
People who predominantly sit down often suffer from spinal complaints. This is mainly caused or intensified by a lack of exercise and a shortened posterior muscle chain.

This study aims to investigate whether CrossFit can improve physical deficits, reduce pain, and improve quality of life.

For this purpose, 30 test persons should take part in regular CrossFit training twice a week over one year. In addition, as a control group, 30 persons are also observed who exercise according to their ideas.

ELIGIBILITY:
Inclusion Criteria:

* Predominantly sedentary work
* Willingness to participate in CrossFit training

Exclusion Criteria:

* Medical reasons against participating in regular exercise
* Acute severe injuries to the musculoskeletal system (e.g. broken bones, torn tendons)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Mobility | 1 year
  Changes in the Functional Movement Screen (FMS) according to Cook G. et al.; Int J Sports Phys Ther, 2014. FMS has a range from 0 -21 (0 = worst, 21 = best).

SECONDARY OUTCOMES:
Strength Symmetry | 1 year
  Strength was assessed in kg using the Dr. WOLFF BackCheck® 617 (BC). The BC allows to measure maximum isometric strength. Furthermore, it provides reference data to evaluate strength and strength symmetry values on a scale ranging from 0 - 10 (0 = worst, 10 = best)
Strength | 1 year
  Strength was assessed in kg using the Dr. WOLFF BackCheck® 617 (BC).
Subjective Well-Being | 1 year
  Subjective Well-Being was measured with the World Health Organization Well-Being Index (WHO-5). WHO-5 has a range from 0 -25 (0 = worst, 25 = best).

CONTACTS AND LOCATIONS:
Overall Officials: Annette Schmidt, Dr., Principal Investigator — Bundeswehr University Munich
Locations (1):
- Universität der Bundeswehr, Neubiberg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided